CLINICAL TRIAL: NCT02665871
Title: Safety Study of Freeze-dried Live Attenuated Influenza Vaccine for Intranasal Administration in Chinese Adults Aged 3 Years and Older
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Beijing Chaoyang District Centre for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: cycdc2015-4
Record Dates: First submitted 2016-01-21; First posted 2016-01-28 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-01

CONDITIONS: Influenza
Keywords: vaccine; safety; intranasal administration
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- one dose of Influenza Vaccine in aged 18 years and older (Experimental): One dose of Freeze-dried Live Attenuated Influenza Vaccine for Intranasal Administration in aged 18 years and older
  Interventions: Biological: one dose of Influenza Vaccine
- One dose of Influenza Vaccine in aged 3-17 year (Experimental): One dose of Freeze-dried Live Attenuated Influenza Vaccine for Intranasal Administration in aged 3-17 years
  Interventions: Biological: one dose of Influenza Vaccine
- placebo in aged 18 years and older (Placebo Comparator): placebo in 10 subjects aged 18 years and older on day 0
  Interventions: Biological: placebo
- placebo in aged 3-17 years (Placebo Comparator): placebo in 10 subjects aged 3-17 years on day 0
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: one dose of Influenza Vaccine
  Arms: one dose of Influenza Vaccine in aged 18 years and older
Biological: one dose of Influenza Vaccine
  Arms: One dose of Influenza Vaccine in aged 3-17 year
Biological: placebo
  Arms: placebo in aged 18 years and older
Biological: placebo
  Arms: placebo in aged 3-17 years

SUMMARY:
This study evaluates the safety of freeze-dried live attenuated influenza vaccine for intranasal administration in chinese adults aged 3 years and older.80 subjects will be divided into 2 groups, including 18 years and older and 3-17 years old. Subjects in each groups will randomly receive one dose of influenza vaccine or placebo in a 3:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects more than 3 years
2. Guardian and/or subjects aged at least 10 subjects can be informed consent, and sign a written Informed Consent Form.
3. Subjects, Guardians and his family can obey the demands of the scheme .
4. Axillary temperature less than 37℃

Exclusion Criteria:

1. Subjects with flu or infected with flu within 3 months.
2. Subjects have a vaccine allergies, allergic to any kind of composition in experimental vaccine, such as eggs, ovalbumin etc.
3. Subjects have serious side effects to vaccine, such as allergy, urticaria, skin eczema, dyspnea, angioneurotic edema or abdominal pain.
4. Subjects have symptoms of acute infection within a week.
5. Subjects have autoimmune disease or immune function defect, Subjects have used immunosuppressive therapy, cytotoxic treatment or inhaled corticosteroids in the past 6 months.
6. Subjects have congenital malformations, developmental disorder or serious chronic diseases( such as Down's syndrome, diabetes, Sickle cell anemia or nerve system disease)
7. Subjects have asthma unstable that need emergency treatment, hospitalization, intubation, oral or intravenous corticosteroid in the past 2 years.
8. Subjects have medical history or family history of convulsions, seizures, encephalopathy and psychiatric disease.
9. Alienia, functional asplenia, and alienia or splenectomy in any situation.
10. Serious neurological disorders such as Green Barry syndrome.
11. Subjects have received blood products or immunoglobulin products within 3 months before experimental vaccine inoculated.
12. Subjects have received other study drug in the past month or received live vaccine, subunit vaccine or inactivated vaccine.
13. The indicators of blood test or urine test do not conform to the inclusion criteria.
14. Subjects have received allergy treatment in in the past 14 days.
15. Subjects are receiving anti-tuberculosis treatment.
16. Subjects have inoculated flu vaccine in the flu reason.
17. Axillary temperature is more than 37℃ before vaccination.
18. Subjects are pregnant or plan to become pregnant
19. Subjects are participate in other clinical trials.
20. Any factors unsuitable for clinical trail at the discretion of the investigator.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the rate of adverse reactions of Live Attenuated Influenza Vaccine for Intranasal Administration | 3 months
  Adverse reactions associated with vaccine will be observed in subjects after vaccination. Solicited local adverse events include Pain, Redness, Swelling, Induration, Rash, Pruritus at injection site. solicited general adverse events include Fever, Nausea, Vomiting, Diarrhea, Decreased appetite, Be agitated (irritability, abnormal crying), fatigue, allergy